CLINICAL TRIAL: NCT04086186
Title: Clinical Outcomes of an Adductor Canal Block Versus Liposomal Bupivacaine in Total Knee Arthroplasty Patients: A Randomized Prospective Study
Brief Title: Adductor Canal Block Versus Liposomal Bupivacaine in TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Good Samaritan Regional Medical Center, Oregon (Other)
Responsible Party: Principal Investigator, Justin Than, Orthopedic Resident, Good Samaritan Regional Medical Center, Oregon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-021
Record Dates: First submitted 2019-03-13; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Total Knee Arthroplasty; Post-operative Pain Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adductor Canal Block Group (Active Comparator): Standard method for peri-operative pain control. Adductor canal block is performed by anesthesiologist prior to surgery.
  Interventions: Procedure: Adductor canal block
- Liposomal Bupivacaine Group (Experimental): Experimental method for peri-operative pain control. Liposomal bupivacaine peri-articular injection is performed by surgeon during surgery.
  Interventions: Procedure: Liposomal Bupivacaine Peri-articular Injection

INTERVENTIONS:
Procedure: Liposomal Bupivacaine Peri-articular Injection — A 20mL solution of 266mg of liposomal bupivacaine (Exparel) was mixed with 40mL of normal saline, which was then infiltrated consistently in the posterior capsule, medial and lateral side of the arthrotomy, patella tendon, quadriceps tendon, quadriceps musculature, and subcutaneous soft tissue.
  Other Names: Exparel peri-articular injection
  Arms: Liposomal Bupivacaine Group
Procedure: Adductor canal block — Anesthesiologist performs preoperative adductor canal block using 15mL of 0.5% Bupivacaine HCl
  Arms: Adductor Canal Block Group

SUMMARY:
This is a randomized prospective study of 60 patients undergoing total knee arthroplasty evaluating the clinical outcomes of liposomal bupivacaine periarticular injections (PAI) when compared to single shot adductor canal block using bupivacaine HCl.

DETAILED DESCRIPTION:
Total knee arthroplasty(TKA) is an effective solution for end stage arthritis of the knee; however, post-surgical pain can be difficult to manage and the optimal peri-operative pain management strategy has not been established. This study serves to evaluate the clinical outcomes of liposomal bupivacaine PAI when compared to single shot adductor canal block using bupivacaine HCl in patients undergoing a TKA. The investigators hypothesized that peri-articular injection with liposomal bupivacaine would not be inferior to an adductor canal block using bupivacaine HCl. A total of 60 patients were recruited. Thirty patients were randomized to receive intraoperative liposomal bupivacaine periarticular injection, and another thirty patients randomized to receive a pre-operative adductor canal block using bupivacaine. Both groups otherwise received standard pain management strategies peri-operatively. The primary outcome of interest was post-operative pain, which was measured using the Visual Analog Scale (VAS). Secondary measures included changes in patient function which was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), knee range of motion, post-operative ambulation distance, and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing unilateral primary total knee arthroplasty for end stage osteoarthritis or rheumatoid arthritis.
2. All adults > 18 years of age.

Exclusion Criteria:

1. Not cleared by PCP and appropriate specialists to undergo TKA (Check No if patient has been cleared.)
2. Adults undergoing bilateral primary total knee arthroplasties.
3. Women who are pregnant.
4. Women who are breastfeeding.
5. Inability to receive successful spinal anesthesia.
6. Allergy to amide anesthetics.
7. Inability to receive IV tranexamic acid.
8. Patients who are unable to speak English.
9. Patients who are less than 66kg.
10. Patients who are opioid dependent. We define opioid dependency as patients who are on a long-acting narcotic or patients who are taking more than six tablets of hydrocodone 5mg or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | VAS pain score on post-operative day #1
  Visual analog pain scale ranges from zero (no pain) to 10 (maximum pain)
Visual Analog Scale (VAS) | VAS pain score on post-operative day #2
  Visual analog pain scale ranges from zero (no pain) to 10 (maximum pain)
Visual Analog Scale (VAS) | VAS pain score on post-operative day #4
  Visual analog pain scale ranges from zero (no pain) to 10 (maximum pain)
Visual Analog Scale (VAS) | VAS pain score on post-operative day #7
  Visual analog pain scale ranges from zero (no pain) to 10 (maximum pain)

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Outcome measure will be assessed up to 8 weeks
  Reported WOMAC Score ranges between 0 (worst) to 100 (best)
Knee range of motion | Outcome measure will be assessed up to 8 weeks
  Knee flexion and extension will be recorded during follow up visits
Ambulation distance after surgery | Recorded on post-operative day #1
  Distance walked in feet will be assessed and recorded by physical therapist
Hospital length of stay | Measure outcome will be assess through study completion, on average of 1 year
  Measured by number of nights patient stayed in hospital after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Justin Than, DO, Principal Investigator — Samaritan Health Services
Locations (1):
- Good Samaritan Regional Medical Center, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data to be available up to 7 years.

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Affas F, Nygards EB, Stiller CO, Wretenberg P, Olofsson C. Pain control after total knee arthroplasty: a randomized trial comparing local infiltration anesthesia and continuous femoral block. Acta Orthop. 2011 Aug;82(4):441-7. doi: 10.3109/17453674.2011.581264. Epub 2011 May 11. PMID 21561303
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Tong YC, Kaye AD, Urman RD. Liposomal bupivacaine and clinical outcomes. Best Pract Res Clin Anaesthesiol. 2014 Mar;28(1):15-27. doi: 10.1016/j.bpa.2014.02.001. Epub 2014 Mar 15. PMID 24815964
- [Background] Maheshwari AV, Blum YC, Shekhar L, Ranawat AS, Ranawat CS. Multimodal pain management after total hip and knee arthroplasty at the Ranawat Orthopaedic Center. Clin Orthop Relat Res. 2009 Jun;467(6):1418-23. doi: 10.1007/s11999-009-0728-7. Epub 2009 Feb 13. PMID 19214642
- [Background] Suarez JC, Al-Mansoori AA, Kanwar S, Semien GA, Villa JM, McNamara CA, Patel PD. Effectiveness of Novel Adjuncts in Pain Management Following Total Knee Arthroplasty: A Randomized Clinical Trial. J Arthroplasty. 2018 Jul;33(7S):S136-S141. doi: 10.1016/j.arth.2018.02.088. Epub 2018 Mar 12. PMID 29628196
- [Background] Zlotnicki JP, Hamlin BR, Plakseychuk AY, Levison TJ, Rothenberger SD, Urish KL. Liposomal Bupivacaine vs Plain Bupivacaine in Periarticular Injection for Control of Pain and Early Motion in Total Knee Arthroplasty: A Randomized, Prospective Study. J Arthroplasty. 2018 Aug;33(8):2460-2464. doi: 10.1016/j.arth.2018.03.014. Epub 2018 Mar 16. PMID 29656977
- [Background] Snyder MA, Scheuerman CM, Gregg JL, Ruhnke CJ, Eten K. Improving total knee arthroplasty perioperative pain management using a periarticular injection with bupivacaine liposomal suspension. Arthroplast Today. 2016 Jan 11;2(1):37-42. doi: 10.1016/j.artd.2015.05.005. eCollection 2016 Mar. PMID 28326395
- [Background] Smith EB, Kazarian GS, Maltenfort MG, Lonner JH, Sharkey PF, Good RP. Periarticular Liposomal Bupivacaine Injection Versus Intra-Articular Bupivacaine Infusion Catheter for Analgesia After Total Knee Arthroplasty: A Double-Blinded, Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Aug 16;99(16):1337-1344. doi: 10.2106/JBJS.16.00571. PMID 28816893
- [Background] Schwarzkopf R, Drexler M, Ma MW, Schultz VM, Le KT, Rutenberg TF, Rinehart JB. Is There a Benefit for Liposomal Bupivacaine Compared to a Traditional Periarticular Injection in Total Knee Arthroplasty Patients With a History of Chronic Opioid Use? J Arthroplasty. 2016 Aug;31(8):1702-5. doi: 10.1016/j.arth.2016.01.037. Epub 2016 Jan 30. PMID 26897490
- [Background] Jain RK, Porat MD, Klingenstein GG, Reid JJ, Post RE, Schoifet SD. The AAHKS Clinical Research Award: Liposomal Bupivacaine and Periarticular Injection Are Not Superior to Single-Shot Intra-articular Injection for Pain Control in Total Knee Arthroplasty. J Arthroplasty. 2016 Sep;31(9 Suppl):22-5. doi: 10.1016/j.arth.2016.03.036. Epub 2016 Mar 26. PMID 27113945
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Yu S, Szulc A, Walton S, Bosco J, Iorio R. Pain Control and Functional Milestones in Total Knee Arthroplasty: Liposomal Bupivacaine versus Femoral Nerve Block. Clin Orthop Relat Res. 2017 Jan;475(1):110-117. doi: 10.1007/s11999-016-4740-4. PMID 26883652
- [Background] Kirkness CS, Asche CV, Ren J, Gordon K, Maurer P, Maurer B, Maurer BT. Assessment of liposome bupivacaine infiltration versus continuous femoral nerve block for postsurgical analgesia following total knee arthroplasty: a retrospective cohort study. Curr Med Res Opin. 2016 Oct;32(10):1727-1733. doi: 10.1080/03007995.2016.1205007. Epub 2016 Jul 18. PMID 27326760
- [Background] Horn BJ, Cien A, Reeves NP, Pathak P, Taunt CJ Jr. Femoral Nerve Block vs Periarticular Bupivacaine Liposome Injection After Primary Total Knee Arthroplasty: Effect on Patient Outcomes. J Am Osteopath Assoc. 2015 Dec;115(12):714-9. doi: 10.7556/jaoa.2015.146. PMID 26618816
- [Background] Cien AJ, Penny PC, Horn BJ, Popovich JM, Taunt CJ. Comparison Between Liposomal Bupivacaine and Femoral Nerve Block in Patients Undergoing Primary Total Knee Arthroplasty. J Surg Orthop Adv. 2015 Winter;24(4):225-9. PMID 26731385
- [Background] Broome CB, Burnikel B. Novel strategies to improve early outcomes following total knee arthroplasty: a case control study of intra articular injection versus femoral nerve block. Int Orthop. 2014 Oct;38(10):2087-9. doi: 10.1007/s00264-014-2392-0. Epub 2014 Jun 18. PMID 24938586
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Saranteas T, Anagnostis G, Paraskeuopoulos T, Koulalis D, Kokkalis Z, Nakou M, Anagnostopoulou S, Kostopanagiotou G. Anatomy and clinical implications of the ultrasound-guided subsartorial saphenous nerve block. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):399-402. doi: 10.1097/AAP.0b013e318220f172. PMID 21697687